CLINICAL TRIAL: NCT05765721
Title: Development of Family-based Frailty Selfmanagement Model and the Effects of the FRAIL-SM Program Among Patients With Heart Failure
Brief Title: Family-based Frailty Self Management Model and the Effects of the FRAIL-SM Program Among Patients With Heart Failure
Acronym: FRAIL-SM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YM111045EF
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Frailty; Quality of Life; Self-management
Keywords: Frailty; Quality of Life; self management; Heart failure; family-based program
MeSH Terms: conditions — Frailty; Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients in the intervention group will receive an 8-week family-based frailty self-management program including:individual consultation, teaching how to do self-management by family-based frailty self-management video.
Who Masked: Outcomes Assessor
Masking Description: Research assistants are trained for being outcomes assessors in this study who did not know the allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Patients in this group will receive a 8-week family-based frailty self-management program including: (1) one 20-30 minute individual consultation (teaching how to join the family-based frailty self-management program by using poster); (2) provided self-management booklet; (3) provided family-based frailty self-management program video through Line group meeting, once per two weeks ; (4) individual consultation through telephone follow-up once per week for 8 weeks
  Interventions: Behavioral: FRAIL-SM Program
- Control group (No Intervention): Patients in this group maintain their daily life activities, and there is no intervention given.

INTERVENTIONS:
Behavioral: FRAIL-SM Program — Patients in experimental group will receive a 8 week family-based frailty self-management program; patients in control group maintain their usual life activities.
  Arms: intervention group

SUMMARY:
This randomized controlled trial study aims to develop a frailty self-management model for heart failure patients, and to examine the effect of family-based frailty self-management program (FRAIL-SM) including Family involvement, self-Regulation, Autonomy support, Information sharing and Linkage on frailty, knowledge, self-care ability and quality of life in patients with heart failure and their family's strain, knowledge, confedence, and quality of life. Data is collected by a structural questionnaire including frailty, heart failure knowledge, self-care of heart failure, anxiety and depression, social support, and quality of life and physical indicators at baseline, 4 weeks, 8 weeks and 12 weeks after enrollment.

DETAILED DESCRIPTION:
This study aims to develop a frailty self-management model for heart failure patients, and to examine the effect of family-based frailty self-management program (FRAIL-SM) including Family involvement, self-Regulation, Autonomy support, Information sharing and Linkage on frailty, self-care ability and quality of life in patients with heart failure and their family's strain and quality of life. Patients are recruited with a convenience sampling from two medical centers in Taiwan.

A cross-sectional study is adopted to examine the associated factors of frailty and self-management in patients with heart failure. Besides, a qualitative research with face-to-face individual interview is conducted to understand the experience of frailty and self-management in patients with heart failure and their families. Then, a randomized controlled trial is conducted. Subjects are selected using a convenience sampling and are randomly assigned to the intervention or control group. Patients in the intervention group will receive an 8-week family-based frailty self-management program. Data is collected by a structural questionnaire including frailty, heart failure knowledge, self-care of heart failure, anxiety and depression, social support, and quality of life and physical indicators such as levels of B-type natriuretic peptide, hemoglobin, hematocrit, albumin at baseline, 4 weeks, 8 weeks and 12 weeks after enrollment. Data analysis includes descriptive statistics, Pearson correlation coefficient, independent t-test, chi-square, one-way ANOVA, multiple regression, structural equation modeling, and generalized estimating equation.

ELIGIBILITY:
Patients Inclusion Criteria:

1. aged ≥ 40 years.
2. diagnosed by doctros with heart failure and in stable condition.
3. clear consciousness, can communicate with Chinese and Taiwanese.
4. consent to join in this study.
5. have a smartphone or computer and be able to join social media
6. have SOF score ≥ 1

Patients Exclusion Criteria:

1. were bed-ridden or unable to perform activities of daily living independently.
2. diagnosed by doctors with cognitive dysfunction, mental illness, or severe depression
3. in the acute stage of the disease, such as inflammation, infection, or vascular embolism
4. with contraindications to exercise, such as those with uncontrolled arrhythmia, unstable heart rate, BP or PaO2.
5. suffer from neurological, muscular, skeletal or rheumatoid diseases that are aggravated by exercise.

Caregivers Inclusion Criteria:

1. aged ≥ 20 years.
2. clear consciousness, can communicate with Chinese and Taiwanese.
3. consent to join in this study with patients.

Caregivers Exclusion Criteria:

1. have serious chronic diseases and need to dependent on others for daily living
2. diagnosed by doctors with cognitive dysfunction, mental illness, or severe depression
3. have an employment relationship with the patient

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Frailty Assessment Scale for Heart Failure( FAS-HF) scores | baseline, 4week, 8week, 12week
  Changes from baseline Frailty Assessment Scale for Heart Failure (FAS-HF) scores including three indicators: physical, Psychological and social , at 4 weeks, 8 weeks, 12 weeks. FAS-HF scale contains 15 items, each item use Likert scale five point scoring, the total scores ranged from 0 to 45,the higher scores indicate higher frailty.
Changes in The Minnesota living with heart failure questionnaire(MLHFQ) scores | baseline, 4week, 8week, 12week
  Changes from baseline Minnesota living with heart failure questionnaire at 4 weeks, 8 weeks, 12 weeks. The Minnesota living with heart failure questionnaire contains 21 questions regarding the effects of heart failure on patients' physical (eight questions),emotional (five questions) and general (eight questions) dimensions. The possible answer for each question ranges from 0(no) to 5(a lot), and the total score range is 0-105; a higher score indicates lower quality of life .
Changes in the Self-Care of Heart Failure Index scores | baseline, 4 weeks, 8 weeks, 12 weeks
  Changes from baseline Self-Care of Heart Failure Index scores including three indicators: self-maintenance, self-management and self confidence , at 4 weeks, 8 weeks, 12 weeks. This scale contains 22 items, each item use Likert scale four point scoring, the total scores ranged from 22 to 88, the higher scores indicate better self-care.

SECONDARY OUTCOMES:
Changes in symptoms distress scores | baseline, 4week, 8week, 12week
  Changes from baseline symptoms distress scores at 4 weeks, 8 weeks, 12 weeks. Symptoms distress scale contains 17 common symptoms items, each item use Likert scale five point scoring, the total scores ranged from 17 to 85, the higher scores indicate worse symptom distress
Changes in anxiety and depression scores | baseline, 4week, 8week, 12week
  Changes from baseline hospital anxiety and depression scale at 4 weeks, 8 weeks, 12 weeks. The hospital anxiety and depression scale contains 14 questions(7 for assess anxiety and 7 for assess depression), each item use Likert scale four point scoring, the total scores ranged from 0 to 21, the higher scores indicate more severe anxiety and depression level.
Changes in caregivers confidence of heart failure self care | baseline, 4week, 8week, 12week
  Changes in the Self-Care of Heart Failure Index (SCHFI) scores of caregivers from baseline to 4weeks, 8weeks, and12 weeks. The SCHFI is a self-report measure comprised of 15 items rated on a 4-point response scale and divided into 3 subscales: self-care maintenance, self-care management, and self-care confidence. Self-care maintenance consists of 5 items assessing adherance to HF self care recommendations. Self-care management consists of 6 items assessing the ability to recognize and deal with HF symptoms. Self-care confidence consists of 4 items assessing the confidence in control and manage HF symptoms.
Changes in The Caregiver Strain Index(CSI) | baseline, 4week, 8week, 12week
  Changes in the Caregiver Strain Index(CSI) scores of caregivers from baseline to 4weeks, 8weeks, and12 weeks. The CSI is a 13-item objective questionaire designed to assess level of stress experienced by the informal caregivers.
Changes in heart failure knowledge of caregivers | baseline, 4week, 8week, 12week
  Changes in Dutch Heart Failure Knowledge Scale (DHFKS) scores of caregivers from baseline to 4weeks, 8weeks, and12 weeks. The DHFKS consists of 15 items assessing HF knowledge: 4 items regarding general HF information, 6 items regarding HF treatment (diet, fluid restrictions and activity) and 5 items assessing symptoms and symptom recognition.
Changes in caregivers' quality of life | baseline, 4week, 8week, 12week
  Changes in the WHO Quality of Life-Brief(WHOQOL-BREF) Taiwan version scores of caregivers from baseline to 4weeks, 8weeks, and12 weeks. The WHOQOL-BREF Taiwan version is a 28-item questionaire rated on a 5-point response scale. It divides quality of life into 4 domains: physical health, psychological, social relationships and environment.

CONTACTS AND LOCATIONS:
Overall Officials: Ai-Fu Chiou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (2):
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No